CLINICAL TRIAL: NCT07362992
Title: Does Topical Use of Tranexamic Acid During a Cesarean Delivery Reduce Intra-surgical Bleeding? A Randomized ,Multi-center Trial
Brief Title: Topical Tranexamic Acid to Reduce Blood Loss During Cesarean Delivery
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Rabin Medical Center (Other); Meir Medical Center (Other); Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Liat Mor, principal investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0191-25-WOMC
Record Dates: First submitted 2025-11-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery; Postpartum Hemorrhage (PPH); Intraoperative Blood Loss; Hemostasis
Keywords: Tranexamic Acid; Topical Tranexamic Acid; Hexakapron; Cesarean Delivery; Cesarean Section; Elective Cesarean; Postpartum Hemorrhage; Intraoperative Bleeding; Blood Loss Prevention; Uterine Closure; Randomized Controlled Trial; Maternal Outcomes
MeSH Terms: conditions — Postpartum Hemorrhage; Blood Loss, Surgical | interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Tranexamic Acid (TXA) Group (Experimental): Participants in this group will receive topical tranexamic acid (TXA) applied directly to the uterine incision during cesarean delivery. After the baby and placenta are delivered, the surgeon will spray a solution containing 500 mg of TXA (one ampule, 5 mL) diluted in 15 mL of normal saline onto the uterine incision before suturing begins. After the first layer of sutures is placed, a second syringe of the same TXA solution will be sprayed before the second layer of closure. All other aspects of the surgical technique and postoperative care will follow standard practice.
  Interventions: Drug: Tranexamic Acid (Topical)
- Placebo (Normal Saline) Group (Placebo Comparator): Participants in this group will receive a placebo solution of normal saline applied in the same manner and at the same time points as in the TXA group. After the baby and placenta are delivered, the surgeon will spray 20 mL of sterile saline onto the uterine incision before closure, and again before completing the second layer of sutures. All other surgical and postoperative procedures will be identical to those in the TXA group.
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Tranexamic Acid (Topical) — This intervention involves topical application of tranexamic acid (TXA) directly to the uterine incision during cesarean delivery, rather than the conventional intravenous route. A solution containing 500 mg of TXA (one ampule, 5 mL) diluted in 15 mL of normal saline is sprayed evenly over the uterine incision surface after placental delivery and before suturing. A second application of the same solution is sprayed before the second layer of uterine closure. This localized, site-directed use is designed to reduce intraoperative bleeding with minimal systemic absorption, distinguishing it from previously studied intravenous TXA regimens.
  Other Names: Hexakapron
  Arms: Topical Tranexamic Acid (TXA) Group
Other: Normal Saline (Placebo) — This comparator intervention involves topical application of sterile normal saline to the uterine incision at the same time points as in the TXA arm - after placental delivery and before each layer of uterine closure. The saline is visually indistinguishable from the TXA solution, ensuring blinding of participants and surgical teams. This placebo control enables a direct comparison to determine whether the topical TXA application provides added benefit in reducing intraoperative bleeding.
  Other Names: NaCl 0.9%
  Arms: Placebo (Normal Saline) Group

SUMMARY:
The goal of this clinical trial is to learn whether applying topical tranexamic acid (TXA) directly to the uterine incision during cesarean delivery can reduce surgical bleeding compared to placebo. The study will include pregnant women aged 18-51 undergoing elective cesarean delivery at term (37 weeks or more).

The main questions it aims to answer are:

* Does topical TXA shorten uterine closure time?
* Does topical TXA reduce the need for additional hemostatic sutures? Researchers will compare women receiving topical TXA to those receiving placebo (normal saline) to see if TXA reduces intraoperative bleeding and improves surgical outcomes.

Participants will:

* Be randomly assigned to receive either topical TXA or placebo during cesarean delivery.
* Have standard surgery and postoperative care identical in both groups.
* Provide routine clinical data, including hemoglobin levels and recovery outcomes, from their medical records.

DETAILED DESCRIPTION:
Cesarean delivery carries a recognized risk of significant intraoperative bleeding despite standard uterotonic use and established surgical techniques. Tranexamic acid (TXA), an antifibrinolytic medication, reduces surgical blood loss when administered intravenously, but little is known about the effectiveness of topical TXA applied directly to the uterine incision during cesarean delivery. Evidence from other surgical fields suggests that topical TXA may reduce bleeding with minimal systemic absorption.

This study is a multi-center, randomized, double-blind, placebo-controlled trial designed to evaluate whether topical TXA decreases intraoperative bleeding during elective cesarean delivery at term. A total of 112 participants will be randomized in a 1:1 ratio to receive either TXA (500 mg diluted in 15 mL saline) or an identical-appearing saline placebo. The study drug is applied by spraying the solution directly onto the uterine incision after placental delivery and before each layer of uterine closure. Randomization will be stratified by site, and allocation will be concealed using sequentially numbered envelopes opened by a scrub nurse.

All cesarean procedures will follow a standardized operative technique to minimize variability. Intraoperative and postoperative data will be collected from medical records, including operative characteristics, perioperative hemoglobin values, use of additional hemostatic measures, length of stay, and maternal or neonatal complications. Safety monitoring will focus on thromboembolic events, allergic reactions, and postoperative infections, with periodic review by an independent safety officer.

This trial aims to determine whether a localized, low-cost antifibrinolytic intervention can improve hemostasis during cesarean delivery and potentially be incorporated into routine surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 51 years
* Singleton pregnancy
* Elective cesarean delivery scheduled at ≥37+0 weeks of gestation
* First or second cesarean delivery only
* Low transverse uterine incision planned
* Double-layer uterine closure using 1-0 Vicryl sutures
* Ability to provide written informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to tranexamic acid (TXA)
* History of bleeding or coagulation disorders
* Previous postpartum hemorrhage
* Placenta previa or placenta accreta spectrum
* Presence of uterine myomas
* Current use of anticoagulant or antiplatelet medications
* Planned or intraoperative conversion to general anesthesia
* Known uterine malformations
* Known bleeding tendency or thromboembolic disease

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Uterine closure time (minutes) | Intraoperative (during the index cesarean delivery)
  Time from placement of the first uterine stitch to completion of the final uterine stitch including any additional hemostatic sutures (In minutes)
Number of additional hemostatic sutures (count) | Intraoperative (during the index cesarean delivery)
  Total number of extra hemostatic stitches needed for bleeding control beyond the routine two-layer uterine closure

SECONDARY OUTCOMES:
Estimated intraoperative blood loss (mL) | Intraoperative (during the index cesarean delivery)
  Blood loss estimated by the operating surgeon during the cesarean delivery, recorded at the end of the procedure using standardized estimation protocols.
Change in hemoglobin levels | 16-24 hours postoperatively
  Difference between preoperative hemoglobin concentration and hemoglobin measured 16-24 hours after surgery, expressed in g/dL.
Need for additional uterotonic agents | Intra-operative to 24 hours postoperative
  Administration of additional uterotonic medications beyond routine prophylactic Oxycontin during surgery and up to 24 postoperative
Need for blood transfusion | within 30 days postoperativly
  Incidence of red blood cell transfusion due to surgical blood loss or postoperative anemia.
Duration of hospital admission (days) | Postoperative within 30 days from delivery
  Number of days from the cesarean delivery to hospital discharge.
Postoperative complications | Up to 30 days after surgery
  Occurrence of any postoperative maternal complications, including fever, endometritis, wound infection, thromboembolic events, or reoperation
Post-discharge emergency department visits or hospital readmissions | Within 30 days postpartum
  Any maternal emergency department visits or readmissions related to the delivery within one month of cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Amichai Rottenstreich, Principal Investigator — Edith Wolfson Medical center
Locations (4):
- Israel (4):
  - Edith Wolfson Medical Center, Holon, Central District
  - Meir medical center, Kfar Saba
  - Rabin medical center, Petah Tikva
  - Kaplan medical center, Rehovot

IPD SHARING:
Plan to Share IPD: No